CLINICAL TRIAL: NCT02424864
Title: 4D PET-CT Imaging in Esophageal Cancer
Brief Title: 4D FDG PET in Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N14FDG; NL45839.031.13 (Registry Identifier: CCMO)
Record Dates: First submitted 2015-03-30; First posted 2015-04-23 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-01

CONDITIONS: Esophageal Cancer
Keywords: 4D PET-CT
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4D PET-CT (Other): Other intervention: 4D PET-CT
  Interventions: Other: 4d PET-CT

INTERVENTIONS:
Other: 4d PET-CT — Patients will be imaged with 4D-CT images in addition to the normal protocol of FDG-CT image acquisition

SUMMARY:
FDG PET-CT image acquisition in the abdominal and thoracic region is influenced by organ motion. Respiratory movement blurs the metabolic signal of the esophageal tumor and lymph nodes. The investigators hypothesize that the metabolic signal obtained with motion compensation results in higher SUV-max values and clearer demarcation of the esophageal tumor and lymph nodes.

DETAILED DESCRIPTION:
Patients will receive a normal 3D FDG PET-CT scan. By participating in this trial, one extra 4D CT scan will be made. For both the PET and the 4D CT acquisition, the patient gets an abdominal belt around the waist to register breathing motion. No extra FDG PET scan is required for this study. The 4D CT scan is the only intervention which increases the radiation dose exposure compared to the standard PET-CT scan. However, in comparison to the expected radiation dose delivered, if a patient will be treated with curative chemoradiotherapy, this increase in radiation dose is negligible and secondary risks due to this intervention are therefore not increased. For patients who are not eligible for curative treatment the extra dose is also not relevant, given the life expectancy of this group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathology proven esophageal cancer or tumor highly suspicious for esophageal cancer
* > 18 years
* Written informed consent

Exclusion Criteria:

* <18 years
* Possibility of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
The estimation of tumor size of the primary esophageal tumor on 4Dvs 3D FDG PET | one year

SECONDARY OUTCOMES:
Measurement of SUV max, SUV mean, and SUV peak in 4D versus 3D images of esophageal cancer and lymph nodes and number of suspected involved lymph nodes | one year
  measurement of the SUV is a composite measurement in each FDG PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Francine Voncken, MD, Principal Investigator — NKI-AvL
Locations (1):
- The Netherlands cancer Institute, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Voncken FEM, Vegt E, van Sandick JW, van Dieren JM, Grootscholten C, Bartels-Rutten A, Takken SL, Sonke JJ, van de Kamer JB, Aleman BMP. Motion-compensated FDG PET/CT for oesophageal cancer. Strahlenther Onkol. 2021 Sep;197(9):791-801. doi: 10.1007/s00066-021-01761-w. Epub 2021 Apr 7. PMID 33825916